CLINICAL TRIAL: NCT06031701
Title: Effects of a Neuro-psychosocial Teleassistance Programme for Children With Neuromuscular Diseases
Brief Title: Neuro-psychosocial Teleassistance for Neuromuscular Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Deusto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Neuro-e-Motion NMD
Record Dates: First submitted 2023-07-13; First posted 2023-09-11 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Social Competence; Self Esteem; Quality of Life; Social Skills; Neuromuscular Diseases
MeSH Terms: conditions — Social Skills; Neuromuscular Diseases

STUDY DESIGN:
Intervention Model Description: Quasi-experimental pretest-posttest design with a non-equivalent wait list control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Neuro-psychosocial intervention with 12 grupal sessions is offered
  Interventions: Behavioral: Neuro-psychosocial teleassistance program
- Control (Experimental): Waiting list control group
  Interventions: Behavioral: Neuro-psychosocial teleassistance program

INTERVENTIONS:
Behavioral: Neuro-psychosocial teleassistance program — The intervention is carried out in groups of 5 participants and is organised in 12 sessions: 1 session per week of 1h duration. The intervention is aimed at strengthening aspects of social cognition, self-esteem, social skills and aims at a reduction of symptomatology and a general improvement of psychological well-being.

SUMMARY:
This is a clinical trial to assess the effect of a neuropsychosocial intervention by means of telecare aimed at children and adolescents aged 7-16 years with neuromuscular diseases. The intervention is carried out in groups of 5 participants and is organised in 12 sessions: 1 session per week of 1h duration. The intervention is aimed at strengthening aspects of social cognition, self-esteem, social skills and aims at a reduction of symptomatology and a general improvement of psychological well-being.

DETAILED DESCRIPTION:
Development of a neuro-psychosocial tele-assistance programme for groups of children and adolescents affected by various neuromuscular diseases, including Duchenne/Becker muscular dystrophy, limb-girdle dystrophy, etc. In this project the variables of interest and intervention include social cognition, quality of life, psychological symptomatology and coping strategies. The aim of this study is to test whether this programme improves the indicators in the mentioned variables.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed with a neuromuscular disease by a specialist
* Being between 7 and 16 years old
* Having signed an informed consent form through their legal guardians prior to participation in the study
* Having Spanish as one of their main languages
* Having access to a computer (with a camera, microphone and speakers integrated) and Internet connection to take part in the videoconferences

Exclusion Criteria:

* Presence of any other diagnosis or sensory deficit that would prevent the application of the tests or hinder the correct performance of the intervention´s activities
* Being illiterate

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Social cognition - Emotion Recognition | 3 months after the intervention
  Affect Recognition subtest of the Social Perception Domain of the NEPSY-II in the Spanish edition (Korkman et al., 2014) measures the capacity to identify emotions (happy, sad, neutral, afraid, irrationally angry, and disgust) in various images of children
Social cognition - Theory of mind - NEPSY-II | 3 months after the intervention
  Theory of Mind subtest of the Social Perception Domain of the NEPSY-II in the Spanish edition (Korkman et al., 2014) assesses figurative language, imitation skills, and the capacity to comprehend the thoughts, ideas, and beliefs of others and it also evaluates a person's capacity to comprehend how emotions relate to the social context.
Social cognition - Theory of mind - Happé's Strange Stories | 3 months after the intervention
  The Happé's Strange Stories Test is a well-known test of ToM (Happé, 1994; Spanish version: Pousa, 2002). In this study, we used the White et al. (2009) version that has eight story-types. This test evaluates participants capacity to comprehend nonliteral meanings through the reading of brief vignettes.
Social cognition - Theory of mind - RMETC | 3 months after the intervention
  The Reading the Mind in the Eyes test Child version (RMETC) (Baron-Cohen et al., 2001; Spanish version: Rueda et al., 2013), is a TOM test that features 28 photos of individuals. The participant's task is to match the picture with one of the four adjectives that best describes the feelings and thoughts of the person in the picture.

SECONDARY OUTCOMES:
Health-related quality of life | 3 months after the intervention
  How an individual's health status impacts their overall well-being and ability to lead a satisfying life
  The perception of HRQoL is assessed in both healthy and chronically ill children using the Spanish version of the Pediatric Quality of Life Inventory (PedsQLTM 4.0) (Varni et al., 2001). We used the self-report questionnaire in this study for three age ranges: 5-7, 8-12, and 13-18. Physical functioning, emotional functioning, social functioning, and academic functioning are the four dimensions covered by the 23-item assessment. The PedsQL 4.0 provides a physical and a psychosocial summary score in addition to a total score. It is answered through a likert scale with 5 response options that are then converted into quantitative scores ranging from 0-100 points, with a higher score being a better HRQoL.
Psychopathology | 3 months after the intervention
  Behavioral and emotional symptoms
  The Child Behavior Checklist for Ages 6-18 (CBCL/6-18) (Achenbach & Rescorla, 2001) is a multiaxial assessment tool for identifying behavioral and emotional issues in children and adolescents that is aligned with the ASEBA (Achenbach System of Empirically Based Assessment). It has 113 items total, broken down into eight scales for the following syndromes: anxious/depressed, withdrawn/depressed, somatic complaints, social problems, thinking problems, attention problems, rule-breaking behavior and aggressive behavior. Scores for internalizing, externalizing, and overall difficulties are also provided by the items.
Coping strategies - EAN | 3 months after the intervention
  Different styles to deal with stressful situations
  Coping Scale for Children (EAN) (Morales-Rodríguez et al., 2012) is a self-report scale assesses coping strategies and is intended for children aged nine to 12 years. In the instrument, four problems related to the family context, health, schoolwork and social relationships are posed. The nine coping strategies assessed are distinguished between problem-focused coping and unproductive coping.
Coping strategies - ACS | 3 months after the intervention
  Different styles to deal with stressful situations
  Adolescent Coping Scales (ACS) (3rd edition) (Frydenberg and Lewis, 2000): assesses different coping strategies in adolescents aged 12-18 years to cope with their problems. The inventory assesses 18 different coping strategies and consists of 80 items, 79 closed-ended and one open-ended. Furthermore, the 18 strategies are classified into three basic coping styles: problem-directed coping, coping in relation to others, and unproductive coping.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Martínez, PhD, Principal Investigator — University of Deusto
Locations (1):
- University of Deusto, Bilbao, Bizkaia, Spain

IPD SHARING:
Plan to Share IPD: Yes
The plan is open for other researchers to contact the principal investigator of the study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data is available from now until 2025.
Access Criteria: The plan is open for other researchers to contact the principal investigator of the study.